CLINICAL TRIAL: NCT05538403
Title: Assessment of AI Performance for the Detection of Bone Fractures in Children Aged Less Than 2 Years Old in Suspected Child Abuse Setting.
Brief Title: AI Performance for the Detection of Bone Fractures in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0224
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Fracture
Keywords: Aged; Radiography; Paediatric imaging; Artificial intelligence; child abuse
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The artificial intelligence (AI) software BoneView (GLEAMER Company, Paris, France) has been designed, tested and validated to detect and locate recent or semi-recent fractures on standard radiographs.

The objective will be to assess the AI performance for the detection of bone fractures in children aged less than 2 years old in suspected child abuse setting.

These patients benefit from a whole body radiography with a double blind reading by a "generalist" radiologist and a radiologist with expertise in child abuse. This readings will be compared with the AI results.

Hypothesis is that AI is effective for child fractures detection and could be of help especially for radiologists who are not experts in child abuse.

ELIGIBILITY:
Inclusion criteria:

* aged less than 2 years old
* whole body radiography performed for suspected child abuse setting
* report available with a double blind reading (generalist radiologist and radiologist with expertise in child abuse)

Exclusion criteria:

* Radiograph not interpretable ( poor quality)
* AI not applicable

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged less than 2 years old in suspected child abuse setting
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of fracture detected by AI on radiographs | 1 day
  Percentage of fracture detected by AI on radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Millet, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC